CLINICAL TRIAL: NCT06097325
Title: Prevalence and Experiences of Impostor Syndrome in Anaesthesiology Residents and Chief Residents
Brief Title: Impostor Syndrome and Burnout in Swiss Residents and Chief Residents Anaesthesiologists
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University Hospital, Geneva (Other)
Collaborators: Prof. Savoldelli Georges Louis (Unknown)
Responsible Party: Principal Investigator, Mia Gisselbaek, Principal investigator, Dr. Mia Gisselbaek M.D., MSc., University Hospital, Geneva
Other Study IDs: 2022-01782
Record Dates: First submitted 2023-09-29; First posted 2023-10-24 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Impostor Phenomenon; Imposter Syndrome; Burnout, Professional; Burnout, Student
Keywords: Impostor Phenomenon; Imposter Syndrome; Education; Burnout; Survey; Qualitative Research
MeSH Terms: conditions — imposter syndrome; Burnout, Professional; Burnout, Psychological

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Residents in Anaesthesiology: The residents in Anaesthesiology (French-speaking part of Switzerland) will be enrolled to both:
  * Fill a cross-sectional online survey
  * Enter a qualitative study from the beginning of their residency at Geneva's university hospital
  Interventions: Diagnostic Test: Clance impostor phenomenon scale; Diagnostic Test: Maslach Burnout Inventory for Medical Professional
- Chief-Residents in Anaesthesiology: Chief-Residents (Board-certified anaesthesiologists after post-graduate training) in French-speaking part of Switzerland will be enrolled to fill a cross-sectional online survey
  Interventions: Diagnostic Test: Clance impostor phenomenon scale; Diagnostic Test: Maslach Burnout Inventory for Medical Professional

INTERVENTIONS:
Diagnostic Test: Clance impostor phenomenon scale — The CIPS will be used as "diagnostic test" in the online survey.
  Other Names: CIPS
Diagnostic Test: Maslach Burnout Inventory for Medical Professional — The MBI-HSS-MP will be used as "diagnostic test" in the online survey.
  Other Names: MBI-HSS-MP

SUMMARY:
Surveys including a demographic chart, the Clance Impostor phenomenon scale (CIPS) and the Malash burnout inventory for medical personnel (MBI-HSS-MP) will be sent to residents and chief-residents in anesthesiology in Latin Switzerland (VD, VS, GE, Ti).

A qualitative study will then explore the experiences and coping strategies of self-doubt and impostor syndrome of junior resident anesthesiologists working at Geneva University Hospital, during their transition from mandatory training in internal medicine to anesthesiology.

DETAILED DESCRIPTION:
The Impostor syndrome (IS), as first described by Clance and Imes, is the "Inability to internalize success and the tendency to attribute success to external causes such as luck, error or knowing the appropriate individuals". Failure to recognize personal or professional success may lead to a sense of fraudulence or impostorism and may have negative consequences for career advancement and well-being. IS has been described among men and women in multiple settings worldwide. A systematic review of IS found that it often co-occurs with depression and anxiety and can lead to poor job performance and burnout.

A number of studies have explored IS among health professionals and its impact on professional performance. Healthcare professionals with heavy workloads and responsibility for patient care may be exposed to errors, feelings of self-doubt, anxiety and guilt. A recent scoping review of IS among physicians and physicians in training showed that low self-esteem, institutional culture and female gender were associated with higher rates of IS, which was itself associated with higher rates of burnout. Experiences of underperformance and inadequate self-assessment in physicians were also linked to self-doubt and feelings of fraudulence. Medical culture itself may encourage such individual blame and perfectionism.

IS has not been well studied within the field of anesthesia. Anesthesia is a technical medical specialization characterized by its high stress level. Anesthesiologists are subject to burnout and drug dependence due to their work-related stress and facilitated access to medications. The responsibilities to care for patient lives during unstable periods brought by the surgical act or medical condition generates a particularly high tension for anesthesiologists.

The purpose of our study is to assess the prevalence of IS and burnout in Swiss anesthesiology residents and chief residents and explore in depth the experiences and coping strategies of junior resident anesthesiologists in one French-speaking Swiss hospital.

This will be done by first conducting a survey including two scales (one that assess Burnout (MBI-HSS MP) and one that assess Impostor Syndrome (CIPS)) and a demographic part to understand which residents and chief-residents are more prone to endure such feelings. The investigators also want to understand if those feelings are linked to a recent transition either in institutions or in role.

The investigators also want to do in-depth interviews with residents in anesthesiology to understand how and in which situations those feelings arise and to uncover which coping strategies they use.

The proposed study corresponds to risk category A, as participants in the study are not exposed to any direct health risk. Nonetheless, psychological support will be available to the participants taking part in the qualitative sub-study, in the event that surveys and interviews arouse difficult emotions.

These results will be used to identify potential strategies to prevent IS and its negative consequences, potentially burnout, among Swiss anesthesiologists. The investigators plan to construct and implement (Test) interventions aimed at medical students and residents to increase knowledge of impostor syndrome and burnout and to give them tools to react to such feelings.

ELIGIBILITY:
Inclusion criteria for the survey:

• Currently working hospitals included in the COMASUL network (COMmission Latine d'engagement pour l'Anesthésie et SUisse Latine : HUG - CHUV - Lugano - Bellinzona - Morges - Nyon - Rennaz - Payerne - Sion - Neuchâtel - Fribourg)

Exclusion criteria for the survey:

* Working outside of the COMASUL network
* Specialized anaesthesiologists who are not currently chief residents.

Inclusion criteria for the in-depth interviews:

• Beginning anesthesiology residency at Geneva University Hospitals (HUG) in either May or November (standard residency starting times, which will be used as recruitment time)

Exclusion criteria for the in-depth interviews:

• Having started the anesthesiology residency at the HUG before the May or November recruitment times, or having previous work experience at the HUG in the anesthesiology department.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Residents and chief residents in anaesthesiology working in Latin Switzerland.
  Residents are currently undergoing post-graduate medical training in Anaesthesiology
  Chief-Residents have completed their residency and are board-certified Anaesthesiologists working in Swiss institutions.
  We estimate a total population of about 140-150 residents and 100-120 chief residents.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-11-03 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Impostor syndrome | 6 months
  Describe the prevalence of and relationship between impostor syndrome in anaesthesiology residents and burnout (other outcome), as well as key socio-demographics.
  A validated score will be used: the Clance impostor phenomenon scale (CIPS) which is a 20 questions on a 5-point Likert scale that investigate feelings about self-assessment of competency, praise, and success. The higher the score, more the participant is prone to impostor syndrome.
Burnout | 6 months
  Describe the prevalence of and relationship between burnout in anaesthesiology residents and impostor syndrome (other outcome), as well as key socio-demographics.
  The MBI-HSS-MP (Maslach Burnout Inventory for medical personnel) will be used. It is a scale that captures three dimensions of burnout (emotional exhaustion, depersonalization and personal accomplishment) and uses a 7-level frequency scale on 22 questions. For the domains of depersonalization and emotional exhaustion, the higher the score, the more the participant is subject to burnout. For the domain of personal accomplishment, the lower the score, the more the participant is subject to burnout.

SECONDARY OUTCOMES:
Coping strategies used by residents regarding impostor syndrome and burnout | 2 years
  Residents in anaesthesiology will take part in a qualitative study on the experience of burnout and impostor syndrome in anesthesiology and the coping strategies they use.
  The qualitative interviews will assess how residents experience impostor syndrome and burnout and gather coping strategies they employ. A description of coping strategies will yield from analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Mia Gisselbaek, MD, Principal Investigator — University Hospital, Geneva
Locations (1):
- Geneva's university hospitals, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bravata DM, Watts SA, Keefer AL, Madhusudhan DK, Taylor KT, Clark DM, Nelson RS, Cokley KO, Hagg HK. Prevalence, Predictors, and Treatment of Impostor Syndrome: a Systematic Review. J Gen Intern Med. 2020 Apr;35(4):1252-1275. doi: 10.1007/s11606-019-05364-1. Epub 2019 Dec 17. PMID 31848865
- [Background] Sirriyeh R, Lawton R, Gardner P, Armitage G. Coping with medical error: a systematic review of papers to assess the effects of involvement in medical errors on healthcare professionals' psychological well-being. Qual Saf Health Care. 2010 Dec;19(6):e43. doi: 10.1136/qshc.2009.035253. Epub 2010 May 31. PMID 20513788
- [Background] Clance PR, Imes SA. The imposter phenomenon in high achieving women: Dynamics and therapeutic intervention. Psychotherapy: Theory, Research & Practice US: Division of Psychotherapy (29), American Psychological Association; 1978; 15: 241-7
- [Background] Rivera N, Feldman EA, Augustin DA, Caceres W, Gans HA, Blankenburg R. Do I Belong Here? Confronting Imposter Syndrome at an Individual, Peer, and Institutional Level in Health Professionals. MedEdPORTAL. 2021 Jul 6;17:11166. doi: 10.15766/mep_2374-8265.11166. eCollection 2021. PMID 34277932
- [Background] Hutchins H, Rainbolt H. What triggers imposter phenomenon among academic faculty? A critical incident study exploring antecedents, coping, and development opportunities. Human Resource Development International 2016; 20: 1-21
- [Background] Neufeld A, Babenko O, Lai H, Svrcek C, Malin G. Why Do We Feel Like Intellectual Frauds? A Self-Determination Theory Perspective on the Impostor Phenomenon in Medical Students. Teach Learn Med. 2023 Apr-May;35(2):180-192. doi: 10.1080/10401334.2022.2056741. Epub 2022 Apr 17. PMID 35435084
- [Background] Liu RQ, Davidson J, Van Hooren TA, Van Koughnett JAM, Jones S, Ott MC. Impostorism and anxiety contribute to burnout among resident physicians. Med Teach. 2022 Jul;44(7):758-764. doi: 10.1080/0142159X.2022.2028751. Epub 2022 Feb 1. PMID 35104192
- [Background] Freeman KJ, Houghton S, Carr SE, Nestel D. Measuring impostor phenomenon in healthcare simulation educators: a validation of the clance impostor phenomenon scale and leary impostorism scale. BMC Med Educ. 2022 Mar 3;22(1):139. doi: 10.1186/s12909-022-03190-4. PMID 35236357
- [Background] Gottlieb M, Chung A, Battaglioli N, Sebok-Syer SS, Kalantari A. Impostor syndrome among physicians and physicians in training: A scoping review. Med Educ. 2020 Feb;54(2):116-124. doi: 10.1111/medu.13956. Epub 2019 Nov 6. PMID 31692028
- [Background] LaDonna KA, Ginsburg S, Watling C. "Rising to the Level of Your Incompetence": What Physicians' Self-Assessment of Their Performance Reveals About the Imposter Syndrome in Medicine. Acad Med. 2018 May;93(5):763-768. doi: 10.1097/ACM.0000000000002046. PMID 29116983
- [Background] Gurman GM, Klein M, Weksler N. Professional stress in anesthesiology: a review. J Clin Monit Comput. 2012 Aug;26(4):329-35. doi: 10.1007/s10877-011-9328-7. Epub 2011 Dec 17. PMID 22180163
- [Background] Maslach Burnout Inventory - Human Services Survey for Medical Personnel (MBI-HSS (MP)) - Assessments, Tests | Mind Garden - Mind Garden [Internet]. [cited 2022 Sep 28]. Available from: https://www.mindgarden.com/315-mbi-human-services-survey-medical-personne
- [Result] Feenstra S, Begeny CT, Ryan MK, Rink FA, Stoker JI, Jordan J. Contextualizing the Impostor "Syndrome". Front Psychol. 2020 Nov 13;11:575024. doi: 10.3389/fpsyg.2020.575024. eCollection 2020. PMID 33312149
- [Derived] Gisselbaek M, Suppan M, Saxena S, Hudelson P, Savoldelli GL. Association of impostor phenomenon and burnout among Swiss residents and junior anaesthesiologists: results of a cross-sectional survey. BMC Anesthesiol. 2025 Feb 22;25(1):98. doi: 10.1186/s12871-025-02957-8. PMID 39987071